CLINICAL TRIAL: NCT01569347
Title: Multicentric Descriptive Cross-sectional Study Evaluating Cocaine Users in Treatment Center
Brief Title: Clinical and Genetic Factors Associated With Psychotic Symptoms Among Cocaine Abusers
Acronym: PSYCHOCOKE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI10027 / AOM 10165; 2011-A00115-36 (Other: Eudra CT)
Record Dates: First submitted 2012-03-16; First posted 2012-04-03 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Cocaine-induced Psychotic Disorder During Intoxication
Keywords: Cocaine; Cocaine-induced psychosis; Genetic; Clinical; Biological
MeSH Terms: interventions — Interviews as Topic; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — * Hair sampling: cocain and metabolit dosage (last 3 months)
  * Blood sampling : plasmatic DBH activity, polymorphisms of several genes (DBH,D2R, DAT, COMT)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Cocaine users: Adults, cocaine users
  Interventions: Other: Interviews; Other: Blood sample; Other: Hair sample

INTERVENTIONS:
Other: Interviews — Interviews
Other: Blood sample — Blood sample
Other: Hair sample — Hair sample

SUMMARY:
The aim of this study is to determine the clinical, genetic and environmental factors associated with the phenotype "severe psychotic symptoms" caused by cocaine.

DETAILED DESCRIPTION:
The second purpose is to include gene x environment interaction and to analyse the factors associated with the presence or the absence of severe psychotic symptoms induced by cocaine.

ELIGIBILITY:
Inclusion criteria:

* Adults, cocaine users, who have signed an informed consent

Exclusion criteria:

* Poor venous condition (for blood samples), specially protected people, non French speaking, people who refuse to sign the consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lifetime cocaine users
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2012-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
causes and protective factors of Cocaine Induced Psychosis CIP | up to one day after taking cocaine
  1. clinical data
  2. biologic data
  3. genetic data

SECONDARY OUTCOMES:
gene, environment interactions associated with CIP | up to one day after taking cocaine
  clinical and genetic data

CONTACTS AND LOCATIONS:
Overall Officials: Florence VORSPAN, MD, MSC, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Espace Murger, Hôpital Fernand Widal, Paris, France

REFERENCES:
- [Result] Vorspan F, Fortias M, Zerdazi el-H, Karsinti E, Bloch V, Lepine JP, Bellivier F, Brousse G, van den Brink W, Derks EM. Self-reported cue-induced physical symptoms of craving as an indicator of cocaine dependence. Am J Addict. 2015 Dec;24(8):740-3. doi: 10.1111/ajad.12303. Epub 2015 Nov 6. PMID 26541796
- [Result] Karsinti E, Jarroir M, Zerdazi el-H, Bloch V, Dupuy G, Belforte B, Coeuru P, Plat A, Deschenau A, Cottencin O, Gay A, Lack P, Pelissier-Alicot AL, Bellivier F, Lepine JP, Brousse G, Vorspan F. Childhood trauma are not associated with the intensity of transient cocaine induced psychotic symptoms. Psychiatry Res. 2015 Aug 30;228(3):941-4. doi: 10.1016/j.psychres.2015.05.065. Epub 2015 Jun 27. PMID 26154812
- [Result] Vorspan F, Brousse G, Bloch V, Bellais L, Romo L, Guillem E, Coeuru P, Lepine JP. Cocaine-induced psychotic symptoms in French cocaine addicts. Psychiatry Res. 2012 Dec 30;200(2-3):1074-6. doi: 10.1016/j.psychres.2012.04.008. Epub 2012 May 1. PMID 22551940
- [Result] Brousse G, Vorspan F, Ksouda K, Bloch V, Peoc'h K, Laplanche JL, Mouly S, Schmidt J, Llorca PM, Lepine JP. Could the inter-individual variability in cocaine-induced psychotic effects influence the development of cocaine addiction? Towards a new pharmacogenetic approach to addictions. Med Hypotheses. 2010 Dec;75(6):600-4. doi: 10.1016/j.mehy.2010.07.043. PMID 20801583
- [Derived] Icick R, Vorspan F, Karsinti E, Ksouda K, Lepine JP, Brousse G, Mouly S, Bellivier F, Bloch V. Gender-specific study of recurrent suicide attempts in outpatients with multiple substance use disorders. J Affect Disord. 2018 Dec 1;241:546-553. doi: 10.1016/j.jad.2018.08.076. Epub 2018 Aug 13. PMID 30153638